CLINICAL TRIAL: NCT00637364
Title: An Open Label, Non-Randomized, Single-Center, Therapeutic Trial Examining the Feasibility, Safety, and Efficacy of FEP-BY02, a High Intensity Focused Ultrasound Tumor Treatment Device, in Patients With Pancreatic Cancer Pain
Brief Title: High Intensity Focused Ultrasound Tumor Treatment for Pancreatic Cancer Pain
Acronym: HIFU Pancreas
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor is not proceeding with USA human trial at this time
Sponsor: CMED HIFU Development Corporation (Industry)
Responsible Party: Joo Ha Hwang, MD, PhD, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEP-BY02-01; WIRB 20071832
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Pain; Pancreatic Adenocarcinoma; Ductal Adenocarcinoma
Keywords: pain; pancreas; pancreatic cancer; pancreatic adenocarcinoma; ductal adenocarcinoma
MeSH Terms: conditions — Pain; Pancreatic Neoplasms | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: High intensity focused ultrasound, HIFU — The FEP-BY02 HIFU system uses extracorporeal generated high intensity ultrasound, focused on a tumor region of interest, to ablate tissue. A stand-alone B-mode ultrasound is used to locate and define the tumor region of interest. Once defined, the acoustic energy is delivered using a large aperture; fixed focus; sparse transducer array. The concentration of acoustic energy may result in thermal and/or mechanical bioeffects including tissue necrosis, apoptosis, and/or disruption (temporary or permanent) of normal cellular function within the targeted volume (such as nerve conduction).
  The FEP-BY02 High Intensity Focused Ultrasound (HIFU) system is intended to ablate ductal adenocarcinoma of the pancreas with ultrasound-guided targeted delivery of focused ultrasound energy to effect thermal and/or mechanical bioeffects leading to ablation (destruction) of the targeted tumor tissue.

SUMMARY:
This is an open-label, non-randomized, single-center, therapeutic trial in patients with AJCC Stage III or IV pancreatic cancer with tumor related abdominal and/or back pain to evaluate the safety of high intensity focused ultrasound therapy using the FEP-BY02 HIFU system for palliation of pancreatic cancer-related pain. Patients meeting all eligibility criteria without any exclusion criteria will be offered an opportunity to participate in the study. After obtaining informed consent a baseline history, physical examination, laboratory studies, and any additional imaging studies needed will be performed.

The major theoretic risk to the patient with this procedure is the development of acute pancreatitis. If acute pancreatitis were to develop, it should become clinically evident by day 3 following HIFU ablation. Therefore, the initial phase of this pilot study is designed to allow a sufficient interval between HIFU treatments to identify whether this theoretic risk will manifest clinically. Previous clinical experience in China suggests that HIFU of pancreatic tumors is safe without risk of developing severe acute pancreatitis.

Patients treated with HIFU will have approximately 15-20% of the tumor volume treated per session. The first 5 patients (feasibility study) will receive their first HIFU treatment followed by a 3-5 day interval for observation.

Following the feasibility study the results will be reviewed with the FDA. If no serious adverse events are encountered, and the FDA agrees with continuing the study, then the next 5 patients will be treated with an interval of 2-3 days between each treatment. If no serious adverse events are encountered in this group, then the next group of 5 patients will be treated at intervals of 1-2 days between each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Histology proven pancreatic ductal adenocarcinoma in the body or tail of the pancreas with a 1 cm margin of tissue to all named vessels and adjacent organs
* AJCC stage III or IV pancreatic cancer based on imaging criteria (endoscopic ultrasound, CT scan, and/or MRI)
* Presence of mid-abdominal pain or back pain (>=4 at its worst on Brief Pain Inventory) in the week prior to baseline evaluation or requiring any dose of opioid narcotic for pain relief
* Pancreatic tumor that can be evaluated by RECIST criteria
* Pancreatic tumor that can be imaged with transabdominal ultrasonography
* Pancreatic tumors with an adequate window for the HIFU beam without intervening air or colon
* No contraindications for CT/PET imaging
* Karnofsky's performance status of 50% or greater
* Life expectancy greater than 3 months
* Normal coagulation profile (INR <1.6; platelet count >50,000)
* American Society of Anesthesiologists (ASA) class =/<2, not including patient's diagnosis of pancreatic carcinoma
* Normal serum uric acid, calcium, potassium, phosphate and creatinine values
* Willingness and ability to complete follow-up interviews for 24 months following the last HIFU treatment

Exclusion Criteria:

* Previous pancreatic surgery or resection
* Have had previous surgery to remove jaundice causing obstruction
* Active malignancy (not including metastases) or history of other primary source of cancer other than pancreas except for basal cell carcinoma or carcinoma-in-situ of the cervix
* Any other disease, condition or surgery which might confound HIFU therapy, including the requirement for the patient to remain still in the supine position for 90 minutes
* Inability to image the pancreatic tumor with ultrasound
* The presence of bone (e.g., ribs) in the path of the HIFU beam
* The presence of colon in the path of the HIFU beam
* Use of aspirin containing or aspirin-analog products, including herbal supplements that may decrease coagulation, within two weeks of first HIFU treatment
* Currently a prisoner
* Currently experiencing an episode of major mental illness (psychosis, major affective disorder, or schizophrenia)
* Pregnancy at time of enrollment, since this would contraindicate HIFU therapy
* Participation in any other investigational drug, biologic or medical device study within the 30 days prior to the study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Safety of the FEP-BY02 HIFU system determined by the frequency and severity of adverse events (AEs) categorized and graded for severity according to the Common Terminology Criteria for Adverse Events, Version 3.0 (CTCAE) | pre treatment, post treatment, 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months, 18 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joo Ha Hwang, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States